CLINICAL TRIAL: NCT00210626
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Assess the Effect of Recombinant Human Erythropoietin (Epoetin Alfa (PROCRIT®)) on Functional Outcomes in Anemic, Critically Ill, Trauma Subjects
Brief Title: Assess Functional Outcomes in Anemic, Critically Ill, Trauma Patients When Taking Epoetin Alfa
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Collaborators: Ortho Biotech Products, L.P. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR003235; LTTO; (Other: Johnson & Johnson Pharmaceutical Research and Development, L.L.C.); Long Term Treatment Outcomes; (Other: Johnson & Johnson Pharmaceutical Research and Development, L.L.C.); PR04-15-001 (Other: Johnson & Johnson Pharmaceutical Research and Development, L.L.C.)
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Results first posted 2009-12-22 (Estimated); Last update posted 2014-04-21 (Estimated); Status verified 2014-04

CONDITIONS: Anemia
Keywords: Anemia, erythropoetin, Epoetin alfa, erythropoetin recombinant, Critical care, critical illness, intensive care
MeSH Terms: conditions — Anemia; Critical Illness | interventions — Epoetin Alfa

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PROCRIT (Active Comparator)
  Interventions: Drug: PROCRIT
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PROCRIT — 40,000 IU/mL/week for max of 12 weeks
  Arms: PROCRIT
Drug: Placebo — 40,000 IU/mL/week for max of 12 weeks
  Arms: Placebo

SUMMARY:
The purpose of this trial is to evaluate the physical function outcomes in anemic, critically ill, trauma subjects treated with epoetin alfa (PROCRIT®) compared to placebo.

DETAILED DESCRIPTION:
The overall study design is based on the assumption that the maximum increase in red blood cells and their effect often does not occur while a subject is in the ICU and acutely ill. The study hypothesis is that a higher hemoglobin (red blood cells) carries more oxygen and delivers oxygen to the tissues. This should increase the ability of the injured subject to tolerate the physical exertion involved in the recuperative process and thus recover earlier than someone with a lower hemoglobin.

One milliliter of a colorless liquid is injected under the subjects skin weekly during their hospital stay and weekly for up to an additional 12 weeks after hospital discharge.

ELIGIBILITY:
Inclusion Criteria:

* ICU admission secondary to a blunt multi-system traumatic injury
* A leg or pelvic fracture must be one of the injuries sustained
* Male or female
* Age between 18 and 55 years
* Hemoglobin <=12g/dL at study entry
* An expected ICU stay >=2 days
* Glascow Coma Scale (GCS) score must be >= 13 at hospital admission or within 24 hours of admission
* Documented ability to function independently prior to this hospitalization as determined by a subject or proxy interview using the Karnofsky Performance scale and having a score >=80
* Subjects (or appropriate legal representative) must sign the informed consent form after the nature of the study has been fully explained
* Female subjects that can become pregnant must use an adequate contraceptive method (e.g., abstinence, intrauterine device, oral contraceptives, barrier device with spermicide, or surgical sterilization) during study
* Subjects must be literate in their native language in order to complete written self-assessments during the post-hospital discharge phase

Exclusion Criteria:

* Acute burns
* Traumatic Brain Injury (TBI) with admission GCS <= 12 and/or spinal cord injury
* Cause of injury secondary to a fall from a standing position
* Trauma victims transferred into the participating institution > 8 hours post injury
* Subjects not expected to survive 12 months given their injuries and/or pre-existing, uncorrectable medical condition
* Chronic renal failure on dialysis
* Significant hematological disease
* All subjects expected to undergo chemotherapy during the course of treatment
* A current diagnosis of uncontrolled hypertension
* New onset seizures (within three months) or seizures not controlled by medication prior to admission
* Gustillo III fracture, open pelvic fracture, traumatic amputation
* Prior history or diagnosis of deep vein thrombosis (DVT), pulmonary embolism (PE), or genetic coagulation abnormality
* Pregnancy or lactation
* Refusal to accept blood transfusion
* Received an experimental drug or used an experimental medical device within 30 days prior to the planned start of treatment
* Treatment with any recombinant human erythropoietin within 30 days prior to enrollment - Known hypersensitivity to human albumin or mammalian cell-derived products or epoetin alfa
* Employees of the investigator or study center with direct involvement in the proposed study or other studies under the direction of that investigator or study center

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 192 (Actual)
Dates: Start 2005-08; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tracy McGowan, Study Director — Janssen Services, LLC
Locations (21):
- United States (21):
  - Birmingham, Alabama
  - Orange, California
  - Santa Barbara, California
  - Denver, Colorado
  - Gainesville, Florida
  - Hollywood, Florida
  - Miami, Florida
  - Maywood, Illinois
  - Springfield, Illinois
  - Indianapolis, Indiana
  - Baltimore, Maryland
  - St Louis, Missouri
  - Las Vegas, Nevada
  - Cincinnati, Ohio
  - Dayton, Ohio
  - Allentown, Pennsylvania
  - Philadelphia, Pennsylvania
  - Memphis, Tennessee
  - El Paso, Texas
  - Norfolk, Virginia
  - Morgantown, West Virginia

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: ITT subjects were all randomized subjects. Three subjects were randomized prior to screening and failed screening. These 3 subjects did not receive any study medication or procedure prior to discontinuation and are not included in the 192 subjects that started the study.
Groups:
- PROCRIT: 40,000 IU/mL/week for maximum of 12 weeks
- Placebo: Placebo given at equivalent volume (1 mL) as Procrit
Period: Overall Study
Arm/Group | PROCRIT | Placebo
Started | 97 | 95
Completed | 49 | 50
Not Completed | 48 | 45
Not completed — Adverse Event | 1 | 2
Not completed — Protocol Violation | 1 | 5
Not completed — Lost to Follow-up | 11 | 11
Not completed — Death | 1 | 0
Not completed — Withdrawal by Subject | 29 | 20
Not completed — Physician Decision | 0 | 2
Not completed — Sponser Request | 1 | 0
Not completed — Other | 4 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PROCRIT | Placebo | Total
Number analyzed (Participants) | 96 | 92 | 188
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 7 | 3 | 10
  Between 18 and 65 years | 89 | 89 | 178
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.2 (10.94) | 33.5 (11.06) | 32.8 (10.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 35 | 67
  Male | 64 | 57 | 121

OUTCOME MEASURES:

1. Primary Outcome: SF-36 PF Score
Description: Average SF-36 (Medical Outcome Survey Short Form) PF (Physical Function) Score post hospital discharge for each subject. Each subjects SF-36 score is the average of all the post hospital discharge scores. The SF-36 score is a patient reported questionaire related to Physical Function base the score can range from 0 to 100. The worst score is 0 and the best possible score is 100.
Time Frame: Hospital Discharge to Post-Hospital Discharge Week 24
Population: ITT (Intent to Treat), The number of subjects analyzed includes all ITT subjects that did not withdraw from the study prior to hospital discharge.
Measure: Mean (Standard Deviation); unit: Units on a scale.
Arm/Group | PROCRIT | Placebo
Number analyzed (Participants) | 85 | 81
Units on a scale. | 27.30 (23.668) | 30.88 (23.522)
Statistical Analysis 1: Comparison: PROCRIT vs Placebo; The null hypothesis is that there is no difference between Procrit and Placebo in average SF-36 Physical Function Scores; Test type: Superiority or Other; p = 0.3807, ANCOVA; Covariate used is Baseline SF-36 PF Score. Baseline SF-36 PF Score was collected prior to the start of Procrit or Placebo treatment

2. Secondary Outcome: Return to Usual Activity (RTUA)
Description: Number of Subjects with Week 24 SF-36 PF Score greater than or equal to their pre-trauma SF-36 PF score. The pre-trauma SF-36 PF score was collected at hosptital discharge and reflects a subjects physical function before they were injured and hospitalized.
Time Frame: Hospital Discharge to Post-Hospital Discharge Week 24
Population: Intention to Treat(ITT)population and completed Week 24 Post-Hospital discharge.
Measure: Number; unit: Participants
Arm/Group | PROCRIT | Placebo
Number analyzed (Participants) | 35 | 37
Participants | 9 | 11
Statistical Analysis 1: Comparison: PROCRIT vs Placebo; Test type: Superiority or Other; p = 0.7038, Chi-squared

ADVERSE EVENTS:
Arm/Group | PROCRIT | Placebo
Serious Adverse Events (participants affected / at risk) | 17/96 | 20/92
Other Adverse Events (participants affected / at risk) | 83/96 | 81/92
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | PROCRIT (N=96) | Placebo (N=92)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Peritoneal Haemorrhage (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 1
Small Intestinal Obstruction (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Wound Necrosis (General disorders) | 1 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 1
Abdominal Sepsis (Infections and infestations) | 1 | 0
Bacteraemia (Infections and infestations) | 1 | 0
Cystitis (Infections and infestations) | 1 | 0
Lung Infection Pseudomonal (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Urinary Tract Infection (Infections and infestations) | 1 | 0
Wound Infection Staphylococcal (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 0 | 1
Endocarditis (Infections and infestations) | 0 | 1
Infected Skin Ulcer (Infections and infestations) | 0 | 1
Lobar Pneumonia (Infections and infestations) | 0 | 1
Localised Infection (Infections and infestations) | 0 | 1
Osteomyelitis (Infections and infestations) | 0 | 1
Postoperative Wound Infection (Infections and infestations) | 0 | 1
Septic Shock (Infections and infestations) | 0 | 1
Staphylococcal Bacteraemia (Infections and infestations) | 0 | 1
Staphylococcal Infection (Infections and infestations) | 0 | 1
Wound Infection (Infections and infestations) | 0 | 1
Haemothorax (Injury, poisoning and procedural complications) | 1 | 0
Implant Tissue Necrosis (Injury, poisoning and procedural complications) | 1 | 0
Joint Dislocation (Injury, poisoning and procedural complications) | 1 | 0
Post Procedural Haemorrhage (Injury, poisoning and procedural complications) | 0 | 2
Anemia Postoperative (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Fracture Displacement (Injury, poisoning and procedural complications) | 0 | 1
Pneumothorax Traumatic (Injury, poisoning and procedural complications) | 0 | 1
Post-Traumatic Pain (Injury, poisoning and procedural complications) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Aseptic necrosis Bone (Musculoskeletal and connective tissue disorders) | 0 | 1
Fracture Nonunion (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Cerebellar Haematona (Nervous system disorders) | 0 | 1
Dysarthria (Nervous system disorders) | 0 | 1
Delirium (Psychiatric disorders) | 0 | 1
Psychotic Disorder (Psychiatric disorders) | 0 | 1
Renal Failure Acute (Renal and urinary disorders) | 1 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1/92 | 1
Laryngeal Disorder (Respiratory, thoracic and mediastinal disorders) | 0/92 | 1
Deep Vein thrombosis (Vascular disorders) | 4 | 4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PROCRIT (N=96) | Placebo (N=92)
Leukocytosis (Blood and lymphatic system disorders) | 2 | 6
Thrombocythaemia (Blood and lymphatic system disorders) | 7 | 8
Tachycardia (Cardiac disorders) | 2 | 5
Constipation (Gastrointestinal disorders) | 32 | 37
Diarrhoea (Gastrointestinal disorders) | 8 | 11
Nausea (Gastrointestinal disorders) | 20 | 26
Vomiting (Gastrointestinal disorders) | 10 | 5
Odema Peripheral (General disorders) | 5 | 10
Pyrexia (General disorders) | 19 | 21
Pneumonia (Infections and infestations) | 12 | 9
Urinary Tract Infection (Infections and infestations) | 13 | 12
Decreased Appetite (Metabolism and nutrition disorders) | 1 | 5
Hypokalemia (Metabolism and nutrition disorders) | 12 | 8
Hyponatraemia (Metabolism and nutrition disorders) | 4 | 5
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 5
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 8 | 9
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 6 | 10
Dizziness (Nervous system disorders) | 5 | 3
Headache (Nervous system disorders) | 6 | 8
Agitation (Psychiatric disorders) | 7 | 4
Anxiety (Psychiatric disorders) | 6 | 10
Depression (Psychiatric disorders) | 7 | 4
Insomnia (Psychiatric disorders) | 26 | 28
Urinary Retention (Renal and urinary disorders) | 5 | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 | 2
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 4 | 6
Decubitus Ulcer (Skin and subcutaneous tissue disorders) | 2 | 6
Pruritus (Skin and subcutaneous tissue disorders) | 6 | 13
Rash (Skin and subcutaneous tissue disorders) | 5 | 5
Deep Vein Thrombosis (Vascular disorders) | 5 | 6

LIMITATIONS AND CAVEATS:
The study was stopped early due to slow enrollment. Four subjects were randomized but withdrew prior to hospital entry and no data were collected

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All information which is supplied by COBS to the investigator & not previously published & any data generated as a result of the study are confidential & remain the sole property of COBS. Investigator will not use the information for other purposes without COBS prior written consent.